CLINICAL TRIAL: NCT06670144
Title: The Associations Between Diet and Rheumatoid Arthritis Risk in the United Kingdom
Brief Title: Diet and Rheumatoid Arthritis Risk in the United Kingdom Women's Cohort
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Darren Greenwood, Senior Lecturer in Biostatistics, University of Leeds
Other Study IDs: fsydo_UKWCS
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Nutrition; Rheumatoid Arthritis; Alcohol consumption; Body Mass Index; Cohort study; Epidemiology; Arthritis, Rheumatoid, Seropositive
MeSH Terms: conditions — Arthritis, Rheumatoid; Alcohol Drinking; Arthritis | interventions — Dietary Patterns; Ethanol; Fruit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- United Kingdom Women's Cohort: United Kingdom Women's Cohort Study. No interventions are to be administered in this observational prospective cohort study.
  Interventions: Other: Dietary pattern; Other: Alcohol intake; Other: Fruit and vegetables intake; Other: Tea consumption; Other: Coffee consumption; Other: Fish intake; Other: Meat intake; Other: Vitamin D intake

INTERVENTIONS:
Other: Dietary pattern — (regular meat-eater, occasional meat-eater, fish-eater, vegetarian, and vegan; Mediterranean diet)
Other: Alcohol intake — (Frequency and intake of beer, wine, sherry, and spirits were collected by asking the number of specified units (pints, glasses or measures) of each type of alcoholic beverage (beer or cider, wine, sherry or fortified wines, and spirits) per week.)
Other: Fruit and vegetables intake — (Intake of fruits, vegetables, fruits and vegetables combined from food frequency questionnaire)
Other: Tea consumption — (Intake of tea from food frequency questionnaire)
Other: Coffee consumption — (Intake of caffeinated coffee and decaffeinated coffee from food frequency questionnaire)
Other: Fish intake — (Intake of fish from food frequency questionnaire)
Other: Meat intake — (Intake of red meat, processed meat, and poultry from food frequency questionnaire)
Other: Vitamin D intake — (Estimated intake of vitamin D, derived from food frequency questionnaire and any recorded supplemental intake)

SUMMARY:
Rheumatoid arthritis (RA) is the most common inflammatory arthritis, affecting around 1% of the UK population. It affects around 400,000 adults and is characterised by synovial inflammation, cartilage and bone damage that requires lifelong treatment and represents a significant burden for both the individual and society. Diet can affect inflammatory status and RA risk, with varying risks for women on specific diets. Low to moderate levels of alcohol consumption may be associated with lower risk of RA, and those who do not consume enough fruit and vegetables could be at a greater risk than those with adequate intakes. Our research aim is to better understand the role of diet in reducing RA risk in United Kingdom women. The research will use existing dietary and lifestyle data from the United Kingdom Women's Cohort Study and hospital records of RA incidence.

DETAILED DESCRIPTION:
Background: Rheumatoid arthritis (RA) is a typical inflammatory arthritic disease that increases morbidity and mortality of cardiovascular diseases worldwide. Previous observational studies have shown potential for risk reduction through dietary factors modification, but associations between most of dietary factors and RA incidence are still uncertain, and evidence in United Kingdom populations is limited. Therefore, this study aims to assess associations between diet and RA incidence in the United Kingdom Women's Cohort.

Research plan and methods: The dietary and lifestyle data from the United Kingdom Women's Cohort, which recruited 35,372 middle-aged women between 1995-1998, will be used. These data were linked to Hospital Episode Statistics to provide data on the incidence of RA in participants.

Cox regression models will be applied to explore potential associations between dietary factors and RA incidence. Dietary factors will be modelled both as categorical and continuous variables so that models can be fit comparing the risk of RA between categories of intakes and per increment increase in exposure intake (linear dose-response). Restricted cubic splines will be used to model non-linear associations for dietary intake of alcohol, fruits, vegetables, tea, and coffee, since previous research has suggested possible non-linear associations for these variables.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 35 - 69 years at time of recruitment
* Able to provide informed consent

Exclusion Criteria:

* Male
* Not a resident of England
* Unable to link dietary and lifestyle data with hospital episode data
* Missing covariate data
* Rheumatoid arthritis records before or on the date of recruitment

Ages: 36 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The UK Women's cohort profile is published here: https://doi.org/10.1093/ije/dyv173
Sampling Method: Probability Sample
Enrollment: 35372 (Actual)
Dates: Start 1995-01-15 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Rheumatoid Arthritis incidence (first) | Time Frame: age when the completed questionnaire was returned (1995-1998) until age at event, death, or end of study period (19 Mar 2019).
  Incidence of first rheumatoid arthritis ascertained from linkage to Hospital Episode Statistics (HES) data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full data access policy for the UK Women's Cohort Study is available via the study website (https://ukwcs.leeds.ac.uk/).
Supporting Information: Study Protocol, ICF
Time Frame: The full data access policy for the UK Women's Cohort Study is available via the study website (https://ukwcs.leeds.ac.uk/).
Access Criteria: The full data access policy for the UK Women's Cohort Study is available via the study website (https://ukwcs.leeds.ac.uk/).
URL: https://ukwcs.leeds.ac.uk/

REFERENCES:
- [Background] Cade JE, Burley VJ, Alwan NA, Hutchinson J, Hancock N, Morris MA, Threapleton DE, Greenwood DC. Cohort Profile: The UK Women's Cohort Study (UKWCS). Int J Epidemiol. 2017 Apr 1;46(2):e11. doi: 10.1093/ije/dyv173. No abstract available. PMID 26430789
- See also: Study website — https://ukwcs.leeds.ac.uk/